CLINICAL TRIAL: NCT05265078
Title: Estimating Risk of Selected Adverse Events in Patients With Von Willebrand Disease Treated With VEYVONDI® (Vonicog Alfa; Recombinant Von Willebrand Factor)
Brief Title: A Study on Estimated Risks of Certain Adverse Events in Adults With Von Willebrand Disease (VWD) Treated With Veyvondi
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-577-4005; EUPAS45617 (Registry Identifier: EUPAS Register)
Record Dates: First submitted 2022-03-02; First posted 2022-03-03 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Von Willebrand Disease (VWD)
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants Diagnosed With VWD: Participants who have been diagnosed with VWD and prescribed VEYVONDI for the approved indications for the index infusion (first eligible VEYVONDI infusion) will be assessed using secondary data obtained from medical records to evaluate the safety of VEYVONDI in real-world clinical practice. All study data will be retrospectively abstracted from medical records by dedicated clinical research staff in partnership with the treating physician. The data window for this study will begin on 01 January 2019 and end one day before site activation at each site.

SUMMARY:
The main aim of this study is to estimate the risks of certain adverse events in adults with Von Willebrand Disease treated with VEYVONDI. No study medicines will be provided to participants in this study.

Data from medical records of participants diagnosed with Von Willebrand Disease and treated with VEYVONDI will be evaluated during this study.

ELIGIBILITY:
Inclusion criteria:

1. Participants with 18 years of age or older
2. Participants with diagnosis of congenital VWD.
3. Participants received VEYVONDI with or without a FVIII concentrate.
4. Participants must have at least 7 days of observation time after the index dose.
5. Provides informed consent, if required, in accordance with local ethical and institutional requirements. All medical record data will be abstracted retrospectively; therefore, an exemption or waiver of informed consent will be sought from all associated independent ethics committees (IECs) and institutional review boards (IRBs).

Exclusion criteria:

1. History of any other coagulation or platelet disorder (including acquired VWD).
2. History of neutralizing antibodies / inhibitors to VWF or FVIII.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have been diagnosed with VWD and were prescribed VEYVONDI in Europe.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Hypersensitivity Reactions | From 01 January 2019 up to one day before site activation at each site (up to approximately 4 years)
  Hypersensitivity reactions are acute events and are considered an adverse events of special interest (AESI) in this study if they occur within 7 days of the infusion (including the day of the initial VEYVONDI infusion).
Percentage of Participants With Thromboembolic Events | From 01 January 2019 up to one day before site activation at each site (up to approximately 4 years)
  Thrombotic events considered as an AESIs if diagnosed during the 30 days after a VEYVONDI infusion. Thromboembolic events include venous thrombosis, arterial thrombosis, pulmonary embolism, and cerebral artery thrombosis.
Percentage of Participants With VWF or Factor VIII (FVIII) Inhibitor Formation | From 01 January 2019 up to one day before site activation at each site (up to approximately 4 years)
  Percentage of participants with VWF or FVIII inhibitor formation will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- MVZ Gerinnungszentrum Hochtaunus, Bad Homburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5a5d9593acfd41fb?idFilter=%5B%22TAK-577-4005%22%5D